CLINICAL TRIAL: NCT06943274
Title: Effects of Standardized Walking Obstacle Course (SWOC) Activities on Balance, Gait and Endurance in Children With Autism Spectrum Disorder
Brief Title: SWOC Activities on Balance, Gait and Endurance in Children With Autism Spectrum Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/RCR/AHS/25/Kainat Subtain
Record Dates: First submitted 2025-04-17; First posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism Spectrum Disorder; Balance; Standardized Obstacle Course; Pediatric balance scale; 6-minute walk test
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial performed, in which 44 children with age of 8-12 years will be taken randomly after meeting inclusion criteria. Children will be divided into two groups. Group A will receive a standard walking obstacle course (e.g balance beam, stepping stones, hurdles, soft mats, gait and endurance activities) 2-3 times a week. Group B will receive other form of physical activities such as standard physical activities (e.g walking, running, climbing, jumping) 2-3 times a week. Pre values were taken at 1st week and post values of intervention will be taken after 4th week of intervention to measure the effects of both therapies.
Who Masked: Participant
Masking Description: The participants were blinded throughout the session but therapist and assessor were not be so it was a single blinded session.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): For Group A Standardized Walking Obstacle Course Activities at least 2-3 times a week during a 4-week period.
  Interventions: Other: Standardized Walking Course Activities
- Group B (Active Comparator): For Group B other physical activities at least 2-3 times a week during a 4-week period.
  Interventions: Other: Common Physical Activities

INTERVENTIONS:
Other: Standardized Walking Course Activities — A randomized controlled trial investigate the effect of a standard walking obstacle course on balance, gait and endurance in children with ASD. Activity could include navigating obstacles of varying height and width balancing on beam, stepping over hurdles and walking on different surfaces.
  * Balance activities
  * Gait activities
  * Endurance activities Start with easier task and end with difficulties. SWOC activities performs 2 to 3 times a week for 4weeks.
  Arms: Group A
Other: Common Physical Activities — Either receive no interventions or engages in a different form of physical activities that doesn't focus on balance gait and endurance e.g standard physical education activities like walking, running, climbing, jumping along with applied behavioral therapy, speech therapy and customized physical therapy.
  Arms: Group B

SUMMARY:
Autism Spectrum Disorder (ASD) is a developmental disorder characterized by challenges in social communication, social interaction, repetitive behaviors, and restrictive interests.

Affecting 0.2-2% of children, ASD often includes motor growth retardation, which worsens over time. The disorder is more commonly diagnosed in boys, and its cause is believed to be genetic, with environmental stimuli potentially activating certain genes. This study aims to explore the effects of Standardized Walking Obstacle Course (SWOC) activities on balance, gait, and endurance in children with ASD, seeking to discover novel treatment techniques that could enhance clinical practices and improve motor skills in these children.

This randomized controlled trial will be conducted over 10 months, with data collected from the Lahore Autism Center and PSRD hospital in Lahore, Punjab. The sample will include 44 children with confirmed ASD, aged 8 to 12 years, divided into two groups: one undergoing SWOC activities and the other receiving conventional physiotherapy. Interventions will occur 4 days a week for 30-40 minutes each day. Pre- and post-treatment measurements will be taken using the Pediatric Balance Scale (PBS), the 6-Minute Walk Test (6MWT), and Functional Gait Assessment (FGA).

Data will be analyzed using SPSS version 24, with statistical significance set at P = 0.05.

DETAILED DESCRIPTION:
4 weeks treatment plan.

Group A: A randomized controlled trial investigate the effect of a standard walking obstacle course activities on balance, gait and endurance in children with ASD. Activity could include navigating obstacles of varying height and width balancing on beam, stepping over hurdles and walking on different surfaces. 2-3 times for 4 weeks. Balance beam Stepping stones Hurdle Markers Soft Mats Balance activities Gait and Endurance activities

Group B: Either receive no interventions or engages in a different form of physical activities that doesn't focus on balance gait and endurance e.g standard physical education activities like walking, running climbing, jumping along with applied behavioral therapy, speech therapy and customized physical therapy. 2-3 times for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Children with confirmed diagnosis of ASD.
* Age of patients 8 to 12 year.
* Both male and female.
* Fall less than 15 times in 30 seconds in Flamingo balance scale test.

Exclusion Criteria:

* Severe physical impairment.
* Severe intellectual impairment.
* Comorbid conditions that could prevent participation.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2025-05-15 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Pediatric Berg's balance scale for balance assessment | Baseline, 4th week
  The Pediatric Balance Scale (PBS), a modification of Berg's Balance Scale, was developed as a balance measure for school-age children with mild to moderate motor impairments.
  Scoring of PBS is from 0 to 56 and more scores means balance is good and less scores indicated poor balance.intraclass correlation coefficient (ICC) model 3,1 = 0.998 or individual items Kappa Coefficients, k = 0.87 to 1.0; Spearman Rank Correlation Coefficients, r = 0.89 to 1.0 (21).
  3.8.2.
6-minute walk test | Baseline, 4th week
  The 6-minute walk test is a submaximal exercise test used to quantify the functional exercise capacity in clinical populations. Test-retest reliability was undertaken in 52 subjects, and the intraclass correlation coefficient (95% confidence interval) was calculated as 0.94 (0.89-0.96).
Gait outcome assessment list | Baseline, 4th week
  Gait outcome assessment is used to measure and analyze an individual's walking ability, commonly employed in clinical settings for rehabilitation assessment or functional evaluation. It involves scoring parameters like speed, stride length, cadence, and balance during walking tests. The Intraclass Correlation Coefficient (ICC) is 0.89.

CONTACTS AND LOCATIONS:
Overall Officials: Kainat Subtain, MS-PPT, Principal Investigator — Riphah International University
Locations (1):
- Rising Sun Institute, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Biffi E, Costantini C, Ceccarelli SB, Cesareo A, Marzocchi GM, Nobile M, Molteni M, Crippa A. Gait Pattern and Motor Performance During Discrete Gait Perturbation in Children With Autism Spectrum Disorders. Front Psychol. 2018 Dec 11;9:2530. doi: 10.3389/fpsyg.2018.02530. eCollection 2018. PMID 30618953
- [Background] Rhiel S, Klay A, Keller U, van Hedel HJA, Ammann-Reiffer C. Comparing Walking-Related Everyday Life Tasks of Children with Gait Disorders in a Virtual Reality Setup With a Physical Setup: Cross-Sectional Noninferiority Study. JMIR Serious Games. 2024 Mar 18;12:e49550. doi: 10.2196/49550. PMID 38498048